CLINICAL TRIAL: NCT01695889
Title: A Case-control Study of Exposure to General Anesthesia and a Diagnosis of Alzheimer´s Disease Later in Life.
Brief Title: Is There a Relationship Between Previous Exposure to General Anesthesia and the Development of Alzheimer´s Disease?
Acronym: DEMA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Anna-Karin Strand, MD, Specialist in Anaesthesiology and Intensive Care, University Hospital, Linkoeping
Other Study IDs: DEMA-1
Record Dates: First submitted 2012-09-27; First posted 2012-09-28 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Alzheimer´s Disease; General Anesthesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare exposure to general anesthesia between cases with a diagnosis of Alzheimer´s disease and controls without diagnosis, through studies of medical records. The investigators wish to explore if there is a relationship between exposure to general anesthesia and the development of Alzheimer´s disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer´s disease
* Previous exposure to anesthesia

Exclusion Criteria:

* Inability to retrieve medical records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases from a regional Alzheimer´s disease record. Matched controls from the national population register.
Sampling Method: Non-Probability Sample
Enrollment: 877 (Actual)
Dates: Start 2012-05; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Exposure to general anesthesia | Up to 20 years in retrospect

SECONDARY OUTCOMES:
Exposure to inhaled anesthetics | Up to 20 years in retrospect

CONTACTS AND LOCATIONS:
Overall Officials: Christina Eintrei, professor, Study Chair — University Hospital Linkoping
Locations (1):
- University Hospital, Linköping, Linkoping, Sweden